CLINICAL TRIAL: NCT00622258
Title: A Phase I Dose Escalation Study of RAD001 Administered in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C1104
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2014-09

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: everolimus; mTOR inhibitor; non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Everolimus

ARMS (1):
- Everolimus (Experimental)
  Interventions: Drug: Everolmus

INTERVENTIONS:
Drug: Everolmus
  Other Names: RAD001

SUMMARY:
This study assesses the tolerability, safety, efficacy and pharmacokinetics of everolimus in Japanese patients. Everolimus is administered orally everyday to adult patients with relapsed or refractory non-Hodgkin's lymphoma who have progressed despite standard therapy or for whom standard systemic therapy dose not exist.

ELIGIBILITY:
Inclusion criteria:

* Patients must have histopathologically confirmed diagnosis of non-Hodgkin's lymphoma
* Patients must have disease that is either relapsed or refractory after at least one prior treatment regimen and must not be eligible for any standard treatments
* Patients must not have received autologous stem cell transplant at least within 12 weeks prior to study treatment. If patients received autologous stem cell transplant more than 12 weeks ago, they must be fully recovered from the side effects of such treatment
* Patients who have not received autologous stem cell transplant must be either ineligible for the treatment or, if eligible, patients must have chosen not to receive stem cell transplant
* Patients must have at least one measurable lesion
* Age above 20 years old
* Performance Status 0, 1, or 2 on Eastern Cooperative Oncology Group (ECOG) scale
* Patients with a life expectancy of at least 12 weeks
* Patients must be willing to provide portion of bone marrow aspirate and biopsy during study

Exclusion criteria:

* Patients with history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Patients with prior allogeneic stem cell transplant
* Patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Patients who have received radiation therapy for ≤ 28 days prior to first study treatment or who have not recovered from side effects of such therapy.
* Patients who have received any other investigational agents ≤28 days prior to the first study treatment
* Patients who have received anti-neoplastic therapy within 28 days (60 days for monoclonal antibody or radioimmunotherapy) prior to the first study treatment or who have not recovered from side effects of such therapy
* Patients who have received treatment with oral or intravenous steroids or any immunosuppressive agents ≤ 28 days prior to the first study treatment
* Patients who have received prior therapy with RAD001 or other mTOR inhibitors
* Patient with prior therapy of > 450 U blomycin
* Patients with an active, bleeding diathesis.
* Treatment with any hematopoietic colony-stimulating growth factors (e.g., G-CSF) ≤ 14 days prior to the first study treatment
* Patients who have an impairment of gastrointestinal function or who have gastrointestinal disease that may significantly alter the absorption of study treatment (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
* Patients with active respiratory (excluding interstitial lung disease), skin, mucosal, renal, neurological, or ocular disorder of grade > 1
* Patients with a history of interstitial lung disease of grade ≥ 1
* Patients with a known history of human immunodeficiency virus seropositivity, hepatitis B or C seropositivity

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of RAD001 in Japanese patients with relapsed or refractory non-Hodgkin's lymphoma | whole study period
To assess the pharmacokinetics in Japanese patients | 1st sycle

SECONDARY OUTCOMES:
To seek preliminary evidence of efficacy in this population | Every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Japan (7):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kyoto

REFERENCES:
- See also: Results for CRAD001C1104 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13003